CLINICAL TRIAL: NCT06003842
Title: The Effect of Kinesio® Tex Application on Pain, Functionality, Sleep Quality and Work Performance in Drivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar73
Record Dates: First submitted 2023-08-11; First posted 2023-08-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain; Back Pain; Occupational Diseases
Keywords: taping; Kinesio® Tex; functionality; work performance
MeSH Terms: conditions — Neck Pain; Back Pain; Occupational Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two different Kinesio® Tex taping techniques were applied to the participants. One of these applications is for the upper trapezius muscle and the other is a taping technique applied to support the correct postural posture and trapezius muscle. Banding was applied bilaterally.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The exercise program to be given to the participants consists of stretching, strengthening and postural exercises for the muscles in the neck-back region. While doing the posture exercises, the participants will be asked to do the exercises in front of the mirror in order to correct the wrong postural posture and to provide relaxation.
  Interventions: Other: exercise
- taping group (Experimental): In addition to the exercises, the Kinesio® Tex taping application will remain on the body for 4 days, and then it will be applied 6 times in total, with a 3-day break.
  Interventions: Other: exercise; Other: taping

INTERVENTIONS:
Other: exercise — Stretching exercises for flexion, extension, lateral flexion and rotation, upper trapezius, levator scapula and pectoralis major muscles will be applied in the maximum range of motion of the cervical region in three planes. To increase the mobility of the thoracic region, exercises for thoracic mobility will be given. Strengthening exercises will focus on the back muscles. The resistance of the exercises will be determined according to the individual capacities and strain levels of the participants, and it will be requested to increase the amount of resistance applied depending on the functional developments. You will be asked to perform the exercises twice a day, with 10 repetitions, for 6 weeks. Participants will be asked to hold the position for 3-5 seconds and return to the starting position while doing the strengthening exercises.
Other: taping — After the Kinesio® Tex application, it will remain in the body for 4 days, and then it will be applied 6 times in total, with a 3-day break. It will be stated that the area to be banded should not contain substances such as cream, hair or oil. Upper Trapeze taping will be performed by applying one end of the Y tape to the upper trapeze and the other end to the lower part of the spina scapula, by affixing the tape to the head of the shoulder while standing upright, and keeping the participant's ear tilted towards the other ear as much as possible. Before attaching the rest of the tape, the participant will be asked to bring the shoulder blades closer together and stand upright. In this position, using a mechanical correction technique along the medial line of the scapula along the spine, the rest of the tape will be adhered as an I tape with 35-50% tension.
  Arms: taping group

SUMMARY:
This study was planned to examine the effect of Kinesio® Tex application on pain, functionality, sleep quality and work performance in drivers experiencing neck-back pain.

DETAILED DESCRIPTION:
50 active drivers will be included in the study. The drivers included in the study will be randomly divided into two groups as exercise group and taping group. The home exercise program will be visually explained to both groups and the exercises will be sent to the participants as video. Kinesio® Tex will also be applied to the banding group. Evaluations will be made before treatment and after 6 weeks of treatment. Within the scope of the evaluation, demographic information of the patients, work experience, daily working time, dominant hand, education information (university / high school), type of vehicle used, habit of leaning elbow on the left window, diseases and drugs used, smoking and alcohol use, given after mutual interview will be obtained by recording the answers. Joint range of motion, manual muscle test, pain severity of the individuals participating in the study with the Visual Analog Scale, neck functionality assessment with the Neck Disability Indicator, back functionality assessment with the Quebec Back-Low Back Pain Disability Scale, sleep quality assessment with the Pittsburgh Sleep Quality Index, work performance assessment To be assessed by the Work Role Functioning Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study Having signed the voluntary consent form.
* Being between the ages of 18-65
* Working in home health services for at least 2 years
* Reporting symptoms of localized pain and discomfort in the neck-back region lasting at least 1 week in the last 12 months

Exclusion Criteria:

* The participant's wish to terminate the study
* Receiving physical therapy for neck-back pain in the last 3 months
* Findings such as pins and needles, numbness and tingling in the upper extremity
* Having an allergy to taping
* Presence of a known specific disease that may cause chronic neck-back pain (nerve root compression, postoperative condition in the neck and shoulder regions, peripheral entrapment neuropathy, cervical spine anomaly, severe neck trauma such as whiplash, malignancy, migraine).
* Alcohol and drug addiction
* Psychological conditions that may cause physical burden and recent major operations
* Presence of a skin disease that will affect the neck and back area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Neck Pain Disability Index Questionnaire | 8 weeks
  The scale includes 10 titles. It includes pain sensitivity, heavy lifting, personal hygiene, reading, sleep, headache, concentration, work, driving, social activities. There are 6 answer options according to the severity of the limitation or pain. Scoring is between 0 and 5. The highest score is 50 and the least is 0. The neck disability level classification according to the total score is as follows 0-4: no restrictions 5-14: mild limitation 15-24: moderate limitation 25-34: severe limitation 34 and up: completely restricted
The Quebec Back Pain Disability Scale (QBPDS) | 8 weeks
  The problems caused by back pain are evaluated with 20 different activities from the scale. Its rating is between 0-5. 0 points are expressed as "not difficult at all" and 5 points are expressed as "it is not possible to do". The total score is obtained by summing the answers given to the 20 activities.
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  In the evaluation of the Pittsburgh Sleep Quality Index, 18 items are included in the scoring. The scale has a total of 7 components: sleep duration, habitual sleep efficiency, subjective sleep quality, sleep delay, sleep disturbance, daytime dysfunction, and sleep medication use. Some of the components consist of a single item, while others consist of groupings of several items. Each item scores between 0-3 and the sum of the scores of the 7 components forms the PSQI score. The total score is between 0-21. A high total score indicates a low sleep quality. A total PSQI score of ≤5 indicates "good sleep quality", and >5 indicates "poor sleep quality".
Work Role Functioning Questionnaire (WRFQ) | 8 weeks
  The scale evaluates the difficulties experienced by people while doing their jobs as a percentage of time. In addition, the questionnaire evaluates the effectiveness of the treatment applied. It has five sub-headings as work program (5 questions), Efficiency (7 questions), Physical (6 questions), Mental (6 questions) and Social status (3 questions). It is a scale with 27 questions in total. This scale assesses how often individuals have had difficulties while doing their jobs in the last four weeks. If the expression defined in the question is not related to the profession of the person, he is asked to mark the option "It is not suitable for my profession".

CONTACTS AND LOCATIONS:
Overall Officials: Hakan ZENGİ, Study Chair — Uskudar University
Locations (1):
- İstanbul Büyükşehir Belediyesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pope MH, Goh KL, Magnusson ML. Spine ergonomics. Annu Rev Biomed Eng. 2002;4:49-68. doi: 10.1146/annurev.bioeng.4.092101.122107. Epub 2002 Mar 22. PMID 12117750
- [Background] Rehn B, Nilsson T, Lundstrom R, Hagberg M, Burstrom L. Neck pain combined with arm pain among professional drivers of forest machines and the association with whole-body vibration exposure. Ergonomics. 2009 Oct;52(10):1240-7. doi: 10.1080/00140130902939889. PMID 19787503
- [Background] Bovenzi M. A prospective cohort study of neck and shoulder pain in professional drivers. Ergonomics. 2015;58(7):1103-16. doi: 10.1080/00140139.2014.935487. Epub 2014 Jul 7. PMID 24998325
- [Background] Chapline JF, Ferguson SA, Lillis RP, Lund AK, Williams AF. Neck pain and head restraint position relative to the driver's head in rear-end collisions. Accid Anal Prev. 2000 Mar;32(2):287-97. doi: 10.1016/s0001-4575(99)00126-8. PMID 10688485
- [Background] Morris D, Jones D, Ryan H, Ryan CG. The clinical effects of Kinesio(R) Tex taping: A systematic review. Physiother Theory Pract. 2013 May;29(4):259-70. doi: 10.3109/09593985.2012.731675. Epub 2012 Oct 22. PMID 23088702